CLINICAL TRIAL: NCT01664871
Title: Characterization of Fluoride and Silver Pharmacokinetics of Diammine Silver Fluoride Applied Topically to Teeth of Adults
Brief Title: Pharmacokinetics of Diammine Silver Fluoride
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Universidad Peruana Cayetano Heredia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UC1110
Record Dates: First submitted 2012-08-10; First posted 2012-08-14 (Estimated); Last update posted 2012-08-14 (Estimated); Status verified 2012-08

CONDITIONS: Fluoride and Silver Pharmacokinetics of DSF Applied Topically to Teeth of Adults. Erythema, Bleeding, White Changes, Ulceration and Pigmentation Were Assessed
MeSH Terms: conditions — Hemorrhage; Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Levels of SIlver and Fluoride in Plasma (Experimental)
  Interventions: Device: DIammine SIlver Fluoride

INTERVENTIONS:
Device: DIammine SIlver Fluoride — Concentrations of Silver and Fluoride in the DSF used for study were 24.9% and 5.5%, respectively Average total weight (calculated volume) of Diammine Silver Fluoride applied was 7.57 mg (6.04 µL), corresponding to a mean application of 0.33 mg Fluoride based on the lot analysis. The mean total amount of Silver applied to the 3 teeth was 1.50 mg.

SUMMARY:
There is growing worldwide interest in the use of diammine silver fluoride (DSF) as a topical agent to treat dentin hypersensitivity and dental caries. It has been available in various formulations for many years, but its safety profile has never been fully characterized.

This preliminary study determined the applied doses (3 teeth treated), maximum serum concentrations, and time to maximum serum concentration for fluoride and silver in 6 adults over 4 h. Fluoride was determined using the indirect diffusion method with a fluoride selective electrode, and silver was determined using inductively coupled plasma-mass spectrometry. The mean amount of DSF solution applied to the 3 teeth was 7.57 mg (6.04 µL).

.

DETAILED DESCRIPTION:
Participants Six healthy volunteers (4 females, mean age 36.2, range 23-52 yr) were recruited among staff members of the Universidad Católica de Santa María, Arequipa, Peru. Participants were taking no medications and had most permanent teeth present. Participants were asked to avoid fish or tea for 12 h before the study and not use fluoridated toothpaste 4 h prior. The Comité de Etica de Investigacion, Universidad Católica de Santa María approved the study and informed consent was obtained.

Study Agent DSF [Ag(NH3)2F, CAS RN 33040-28-7, Saforide, Toyo Seiyaku Kasei Co. Ltd. Osaka, Japan] was used. DSF is clear and colorless, with a weak odor of ammonia. The 38% solution contains between 24.4-28.8% (w/v) silver (Ag), and 5.0-5.9% fluoride (F). Concentrations of Ag and F in the DSF used for study were 24.9% and 5.5%, respectively, and the specific gravity was 1.253 at 25°C (Certificate of Analysis Lot #155060). Diammine silver fluoride is also referred to in the literature as silver diammine fluoride, silver diamine fluoride or silver fluoride.

Procedures Three maxillary teeth (cuspid and premolars) in the same quadrant were treated. Three teeth were treated because this was the average number of sensitive teeth reported in an epidemiological study of adults [5]. The teeth were free of restorations or cavitation. The facial surface was dried with cotton gauze and then DSF was applied to the cervical area of each tooth. The teeth were isolated in order to avoid wetting the brush with saliva. Each tooth was coated using a separate microbrush, which was dipped in the DSF and weighed before and after the application (Model S2000, Kern & Sohn GmbH, Balingen, Germany). The sum of the differences in weight of material applied was calculated for each participant.

Blood Collection Immediately before application of DSF and then again at approximately 30 min, 1, 2,3 and 4 h after application, blood was obtained from a peripheral vein. The time periods were picked based on a previous pharmacokinetics study of fluoride varnish [6]. The blood was transferred to a fluoride-free plastic Vacutainer tube with clot activator (BD Vacutainer Plus Plastic Serum Tube, BD Diagnostics, New Jersey). The tubes were spun at 1100 g for 10 min and serum transferred by plastic pipette to plastic cryogenic tubes. The samples were frozen and transported to the University of Washington for analysis.

Analysis Fluoride. Samples were thawed and analyzed in duplicate or triplicate using the diffusion and detection method with hexamethyldisiloxane (HMDS) and Orion F-sensitive electrode [7-8]. To improve detection, the pre-diffusion step was omitted [9], and seals were completed before mixing 1 mL serum with 1 mL HMDS, saturated 3 M H2SO4 [10]. The trapping solution was 20 µmoles 1 M NaOH. It was dried down to eliminate variability of evaporation and residual HMDS before adding 100 µL 3 M acetic acid to a final pH 3.4. Standards were 10 and 100 µM fluoride in the same final concentration of NaOH and acetic acid corresponding to 1 and 10 µM F in the samples. ORION F and sleeve type reference electrodes were coupled with an Accumet Basic 0.1 mV meter (Thermo Fisher Scientific, Milwaukee WI).

Vacutainers were tested for fluoride by adding bovine plasma to 2 tubes and letting them sit overnight before combining the 2 samples and comparing them to plasma directly placed in diffusion dishes. Average concentrations (μM±SD) were 0.34±0.014 and 0.32±0.012, respectively. Therefore, less than 2% F in the serum samples came from the Vacutainers and clot enhancer. Recovery (mean±SD) of 1 nmole/ml F added to bovine serum was 101±4%. Fluoride levels were averaged and are expressed as µM.

Silver. Samples were thawed and analyzed using Inductively Coupled Plasma-Mass Spectrometry (EPA 6020a Rev.1 2007). Serum (0.5 mL) was brought to 2 mL with dilute acid (final concentration: 2% HCl, 1% HNO3; trace metal grade, Fisher, Fairlawn, NJ). Samples were centrifuged (1290 g) for 10 min and filtered (0.45 µm, PTFE; all polypropylene syringe) into 15 mL polypropylene centrifuge tubes. The samples were analyzed on an Agilent 7500CE (Santa Clara, CA) inductively-coupled mass spectrometer (ICPMS) with He as the collision cell gas and an ASX-510 autosampler (CETAC, Omaha, NB). A Micromist nebulizer (Glass Expansion, Pocasset, MA) was used (1.15 L/min carrier gas; no makeup gas). Spray chamber temperature was 2°C. RF power was 1500 W. Ag was quantified using Y as internal standard. Calibrants were diluted with 2% HCl and 1% HNO3 prepared from commercial ICPMS grade solutions (Ultra Scientific, N. Kingstown, RI; BDH Aristar, VWR, Radnor, PA) and ranged from 0.5-50 ng/mL. Calibration was by weighted (1/cps) linear regression. Data was corrected by procedure blank. Values of silver less than 2 ng/mL were recoded to 2. Silver concentrations are expressed as ng/mL.

Soft Tissue Assessment The gingiva adjacent to the application of DSF and the mucosa generally were observed at baseline and 24 h after treatment. Erythema, bleeding, white changes, ulceration and pigmentation were assessed using methods developed for an earlier study [1].

ELIGIBILITY:
Inclusion Criteria:

* Subjects with dental abfraction, erosion or root caries at least in one upper or lower premolar or molar
* Those teeth should have hypersensitivity with cold air

Exclusion Criteria:

* Use of any type of hypersensitivity toothpaste
* Use of pain medication
* Pregnant women
* Individuals with sensitivity to silver or other metal ions

Ages: 10 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2011-07; Primary Completion 2011-08 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Level of Fluoride in Plasma | baseline, 30 minutes, 1 hour, 2 hours, 3 hours, 4 hours
  Samples were thawed and analyzed in duplicate or triplicate using the diffusion and detection method with hexamethyldisiloxane (HMDS) and Orion F-sensitive electrode
Level of Silver in Plasma | baseline, 30 minutes, 1 hour, 2 hours, 3 hours, 4 hours
  Samples were thawed and analyzed using Inductively Coupled Plasma-Mass Spectrometry

SECONDARY OUTCOMES:
Gingival alterations | baseline, immediately after treatment, 24 hours after treatment
  The gingiva adjacent to the application of DSF and the mucosa generally were observed at baseline and 24 h after treatment. Erythema, bleeding, white changes, ulceration and pigmentation were assessed using methods developed for an earlier study

CONTACTS AND LOCATIONS:
Overall Officials: Peter Milgrom, DDS, Principal Investigator — University of Washington; Elsa Vasquez, DDS, Study Director — Universidad Catolica Santa Maria Arequipa; Jorge Castillo, DDS MSD PhD, Study Chair — Universidad Peruana Cayetano Heredia
Locations (1):
- Universidad Catolica Santa Maria, Arequipa, Peru

REFERENCES:
- [Derived] Vasquez E, Zegarra G, Chirinos E, Castillo JL, Taves DR, Watson GE, Dills R, Mancl LL, Milgrom P. Short term serum pharmacokinetics of diammine silver fluoride after oral application. BMC Oral Health. 2012 Dec 31;12:60. doi: 10.1186/1472-6831-12-60. PMID 23272643